CLINICAL TRIAL: NCT01433510
Title: Observational National Clinical Trial of Safety and Tolerance in Patients Suffering of an Allergic Grass Pollen Rhinitis and Treated by Grazax in Real Life Settings
Brief Title: Tolerability of Grazax in Patients With Hayfever in Real Life Settings
Acronym: GRAAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT-15; 2007-003772-20 (EudraCT Number)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic; Rhinoconjunctivitis; Immunotherapy
MeSH Terms: interventions — Grazax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Grazax Tablets 75000 SQT (Experimental): Timothy Extract
  Interventions: Drug: Grazax

INTERVENTIONS:
Drug: Grazax — 1 tablet/day - pre and co-seasonal

SUMMARY:
The purpose of this study is to assess the safety profile of specific immunotherapy with Grazax for three consecutive grass pollen seasons.

DETAILED DESCRIPTION:
To assess the safety profile with Grazax according to the presence or not of polysensitization and/or asthma at enrollment

ELIGIBILITY:
Inclusion Criteria:

* History of grass pollen allergy
* Positive skin prick-test and/or positive specific IgE to grass

Exclusion Criteria:

* Severe, unstable or uncontrolled asthma (FEV1<70% of predicted value)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events related to Grazax | From November 2007 to October 2010 (3 years)
  All adverse events were reported according to the MedDRA dictionary

CONTACTS AND LOCATIONS:
Overall Officials: François FW Wessel, MD, Principal Investigator — Centre Hospitalier Universitaire F-44000 Nantes
Locations (1):
- Centre Hospitalier Universitaire, Nantes, France

REFERENCES:
- [Derived] Wessel F, Chartier A, Meunier JP, Magnan A. Safety and tolerability of an SQ-standardized GRAss ALlergy immunotherapy tablet (GRAZAX(R)) in a real-life setting for three consecutive seasons - the GRAAL trial. Clin Drug Investig. 2012 Jul 1;32(7):451-63. doi: 10.2165/11634270-000000000-00000. PMID 22594491